CLINICAL TRIAL: NCT02693262
Title: Rate Response With CLS Versus Accelerometer and Effect on Both Subjective Symptoms and Objective Outcomes in a Heart Failure Population Implanted With Cardiac Resynchronization With Defibrillator Device: The CLASS Trial
Brief Title: Comparing Rate Response With CLS Versus Accelerometer ICD Settings in Heart Failure Patients With BIOTRONIK CRT-Ds
Acronym: CLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Hsu, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 151774
Record Dates: First submitted 2015-12-24; First posted 2016-02-26 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure; ICD; Chronotropic Incompetence
Keywords: defibrillator; heart failure; ICD; CRT-D; cardiac resynchronization therapy; rate response; CLS; closed-loop stimulation; accelerometer; chronotropic incompetence
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLS Mode on Biotronik CRT-D (Experimental): All 15 patients will be randomized to this group. Their device will be set in the CLS mode for 1 week.
  Interventions: Device: CLS Mode on Biotronik CRT-D
- Accelerometer Mode on Biotronik CRT-D (Active Comparator): All 15 patients will be randomized to this group. Their device will be set in the accelerometer rate responsive mode for 1 week.
  Interventions: Device: Accelerometer Mode on Biotronik CRT-D

INTERVENTIONS:
Device: CLS Mode on Biotronik CRT-D — Setting changed and monitored. Quality of life evaluated through CPET, 6 Minute Walk Test, and Rand 36 Questionnaire.
  Arms: CLS Mode on Biotronik CRT-D
Device: Accelerometer Mode on Biotronik CRT-D — Setting changed and monitored. Quality of life evaluated through CPET, 6 Minute Walk Test, and Rand 36 Questionnaire.
  Arms: Accelerometer Mode on Biotronik CRT-D

SUMMARY:
Dr. Jonathan Hsu and Dr. Eric Adler are conducting a research study to find out more about how implantable cardiac defibrillator (ICD) settings can be adjusted to improve patient cardiovascular health and quality of life. Patients are being asked to participate in this study if they have a history of heart failure and have or are scheduled to be implanted with a BIOTRONIK ICD that is capable of closed loop stimulation (CLS). CLS is a device setting that works with the cardiovascular system to optimize their heart rate during physical activity. This study is comparing BIOTRONIK's CLS setting to a standard accelerometer setting, which also is able to adjust the heart rate by movement sensors, when necessary. This study has been initiated by Dr. Hsu and Dr. Adler and is financially supported by BIOTRONIK, Inc. There will be approximately 15 participants in this trial.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-blind crossover study intended to enroll patients who are implanted or are scheduled to be implanted with a Biotronik CLS and accelerometer capable CRT-D device. Patients will serve as their own control group with regard to modes of rate-adaptive pacing. Patients with a previously implanted Biotronik CRT-D device with CLS-capability will be recruited from health care institutions in San Diego and all dedicated functional testing will be performed at the University of California, San Diego (UCSD). The goal enrollment target for analysis will be 15 patients, with up to 20 patients enrolled to allow for withdrawals.

The purpose of this study is to evaluate whether changes to an implanted ICD can improve the functional status of patients with suspected chronotropic incompetence (CI). CI is a condition in which the heart rate is unable to adequately respond to meet the patient's physical demands, such as walking, climbing stairs, or doing household chores. CI is common in patients with cardiovascular disease, particularly in patients with heart failure. Common clinical management of patients with suspected CI is to activate an accelerometer setting in the cardiac resynchronization therapy with defibrillator (CRT-D) device. An accelerometer will adjust the heart rate to fit the physiological circumstances and needs of the patient based on patient movement only. BIOTRONIK is a company that has developed a novel technology included in the settings for CRT-D devices that offers CLS as an alternative to a standard accelerometer. CLS utilizes sensed electrical properties of the heart in order to assess what may be the best heart rate for both physical and mental demands. This study is designed to compare whether patients will benefit from CLS when compared with standard accelerometer technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BIOTRONIK CRT-D device (capable of CLS and accelerometer rate responsive pacing)
* Patients at least 18 years old
* Patients who have plausible symptoms of CI based on previous monitoring and clinical symptoms

Exclusion Criteria:

* Pregnant patients
* Patients who are unwilling/unable to provide informed consent
* Patients who are unable to complete study related procedures
* Current persistent atrial fibrillation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hsu, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alt E. What is the ideal rate-adaptive sensor for patients with implantable cardioverter defibrillators: lessons from cardiac pacing. Am J Cardiol. 1999 Mar 11;83(5B):17D-23D. doi: 10.1016/s0002-9149(98)01038-8. PMID 10089835
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Faxon DP, Halperin JL, Hiratzka LF, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices); American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices): developed in collaboration with the American Association for Thoracic Surgery and Society of Thoracic Surgeons. Circulation. 2008 May 27;117(21):e350-408. doi: 10.1161/CIRCUALTIONAHA.108.189742. Epub 2008 May 15. No abstract available. PMID 18483207
- [Background] Freedman RA, Hopper DL, Mah J, Hummel J, Wilkoff BL. Assessment of pacemaker chronotropic response: implementation of the Wilkoff mathematical model. Pacing Clin Electrophysiol. 2001 Dec;24(12):1748-54. doi: 10.1046/j.1460-9592.2001.01748.x. PMID 11817808
- [Background] Maass AH, Buck S, Nieuwland W, Brugemann J, van Veldhuisen DJ, Van Gelder IC. Importance of heart rate during exercise for response to cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2009 Jul;20(7):773-80. doi: 10.1111/j.1540-8167.2008.01422.x. Epub 2009 Feb 2. PMID 19207785
- [Background] Coenen M, Malinowski K, Spitzer W, Schuchert A, Schmitz D, Anelli-Monti M, Maier SK, Estlinbaum W, Bauer A, Muehling H, Kalscheur F, Puerner K, Boergel J, Osswald S. Closed loop stimulation and accelerometer-based rate adaptation: results of the PROVIDE study. Europace. 2008 Mar;10(3):327-33. doi: 10.1093/europace/eun024. Epub 2008 Feb 13. PMID 18272507
- [Background] Tse HF, Siu CW, Lee KL, Fan K, Chan HW, Tang MO, Tsang V, Lee SW, Lau CP. The incremental benefit of rate-adaptive pacing on exercise performance during cardiac resynchronization therapy. J Am Coll Cardiol. 2005 Dec 20;46(12):2292-7. doi: 10.1016/j.jacc.2005.02.097. PMID 16360061
- [Background] Keteyian SJ, Isaac D, Thadani U, Roy BA, Bensimhon DR, McKelvie R, Russell SD, Hellkamp AS, Kraus WE; HF-ACTION Investigators. Safety of symptom-limited cardiopulmonary exercise testing in patients with chronic heart failure due to severe left ventricular systolic dysfunction. Am Heart J. 2009 Oct;158(4 Suppl):S72-7. doi: 10.1016/j.ahj.2009.07.014. PMID 19782792
- [Derived] Hsu JC, Darden D, Alegre M, Birgersdotter-Green U, Feld GK, Hoffmayer KS, Han F, Krummen D, Raissi F, Ho G, Taub PR, Urey MA, Adler E. Effect of closed loop stimulation versus accelerometer on outcomes with cardiac resynchronization therapy: the CLASS trial. J Interv Card Electrophysiol. 2021 Sep;61(3):479-485. doi: 10.1007/s10840-020-00829-4. Epub 2020 Aug 5. PMID 32757086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with HFrEF and CI implanted with a CRT-D capable of CLS programming at UCSD were eligible for this study. 102 patients were screened.
Pre-assignment Details: 12 patients signed consent form. 3 participants dropped out of study prior to randomization. 9 participants were randomized and completed study.
Groups:
- CLS, Then DDDR: Participants' CRT devices were initially programmed to no rate response (DDD mode) for a 1-week wash-out period and then were programmed to 1 week of CLS followed by 1 week of DDDR.
- DDDR, Then CLS: Participants' CRT devices were initially programmed to no rate response (DDD mode) for a 1-week wash-out period and then were programmed to 1 week of DDDR followed by 1 week of CLS.
Period: Overall Study
Arm/Group | CLS, Then DDDR | DDDR, Then CLS
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all interventions, therefore baseline characteristics will be reported together.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 69 [63.5 to 76.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Distance (6MWD) Test
Description: Cardiovascular health benefits were measured by the six-minute walk distance (6MWD) test. The 6MWD is a standardized field test to evaluate functional exercise performance. Subjects are instructed to walk as far as possible in 6 min on a flat surface.
  This test was performed twice, once at the end of each intervention period.
Time Frame: Measured on day 14 and day 21.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- CLS Mode on Biotronik CRT-D: All 9 patients will be randomized to this group. Their device will be set in the CLS mode for 1 week.
  CLS Mode on Biotronik CRT-D: Setting changed and monitored. Quality of life evaluated through CPET, 6 Minute Walk Test, and Rand 36 Questionnaire.
- Accelerometer Mode on Biotronik CRT-D: All 9 patients will be randomized to this group. Their device will be set in the accelerometer rate responsive mode for 1 week.
  Accelerometer Mode on Biotronik CRT-D: Setting changed and monitored. Quality of life evaluated through CPET, 6 Minute Walk Test, and Rand 36 Questionnaire.
Arm/Group | CLS Mode on Biotronik CRT-D | Accelerometer Mode on Biotronik CRT-D
Number analyzed (Participants) | 9 | 9
meters | 293.1 (90.2) | 315.1 (95.5)

2. Primary Outcome: RAND-36 Questionnaire
Description: Quality of life of subjects was measured by the RAND-36 which is a generic 36-item questionnaire that measures eight health-related domains stratified by physical health (physical functioning, role limitations due to physical health, pain, and general health) and emotional health (vitality, role limitations due to emotional problems, social functioning, and mental health). Each scale is directly transformed into a 0-100 scale for a total score range of 0-800. Higher scores represent a more favorable health status.
  This test was performed twice, once at the end of each intervention period.
Time Frame: Performed on day 14 and day 21.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLS Mode on Biotronik CRT-D | Accelerometer Mode on Biotronik CRT-D
Number analyzed (Participants) | 9 | 9
score on a scale | 550.8 (123.9) | 489.3 (164.9)

3. Primary Outcome: Cardiopulmonary Exercise Testing (CPET)
Description: Cardiovascular health benefits were determined by measuring the peak heart rate (HR) during Cardiopulmonary exercise testing (CPET). The CPET is performed on a standard treadmill according to the Naughton protocol. During the test, patients inspired room air through a low-resistance mask, and expired oxygen and carbon dioxide partial pressures were measured with a gas analyzer. HR was recorded every 30 seconds during exercise. All patients were encouraged to exercise to maximal effort.
  This test was performed twice, once at the end of each intervention period.
Time Frame: Performed on day 14 and day 21.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CLS Mode on Biotronik CRT-D | Accelerometer Mode on Biotronik CRT-D
Number analyzed (Participants) | 9 | 9
beats per minute | 110.7 (14.7) | 109.7 (14.1)

4. Primary Outcome: Patient Preference
Description: At the end of the study, patients were asked about personal preference regarding CLS over DDDR.
Time Frame: Performed on day 21.
Measure: Count of Participants; unit: Participants
Arm/Group | CLS Mode on Biotronik CRT-D | Accelerometer Mode on Biotronik CRT-D
Number analyzed (Participants) | 9 | 9
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Patients were followed during the whole 3 week study period for any adverse events, assessed on day 0, day 7, day 14 and day 21.
Arm/Group | CLS Mode on Biotronik CRT-D | Accelerometer Mode on Biotronik CRT-D
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT02693262/Prot_SAP_000.pdf